CLINICAL TRIAL: NCT00179036
Title: Biomagnetic Signals of Intestinal Ischemia II
Acronym: SQUID
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alan Bradshaw, Research Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 060426; R01DK058197 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Ischemia
Keywords: Blood supply; Mesentery
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Good blood flow: Group without any ischemia to the small intestine
- Poor blood flow: Group with partial ischemia to the small intestine

SUMMARY:
The lack of blood flow to the small intestine causes mesenteric ischemia. Using a Superconducting QUantum Interference Device (SQUID) which measures the magnetic field of the small intestine, we are hoping to identify abnormalities without surgical intervention.

DETAILED DESCRIPTION:
The electrical activity of the small intestine may contain important information that will help us diagnose gastrointestinal diseases. The major impediment to reducing mortality of mesenteric ischemia is the lack of a noninvasive diagnostic test that identifies the syndrome before extensive necrosis occurs. Mesenteric ischemia is caused by the lack of blood flow to the intestine. The Superconducting QUantum Interference Device (SQUID) measures the magnetic field of the intestinal smooth muscle. By comparing normal smooth muscle and that of patients with mesenteric ischemia, the investigators hope to identify abnormal disease states without surgery.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects and those with diagnosed mesenteric ischemia

Exclusion Criteria:

* Subjects who report a tendency toward claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2000-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To observe a difference in the magnetic activity between the normal and diseased smooth muscle of the small intestine | 2010

SECONDARY OUTCOMES:
Create mathematical and computer models of electrical activity of smooth muscle | 2010

CONTACTS AND LOCATIONS:
Overall Officials: William O. Richards, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Somarajan S, Muszynski ND, Cheng LK, Bradshaw LA, Naslund TC, Richards WO. Noninvasive biomagnetic detection of intestinal slow wave dysrhythmias in chronic mesenteric ischemia. Am J Physiol Gastrointest Liver Physiol. 2015 Jul 1;309(1):G52-8. doi: 10.1152/ajpgi.00466.2014. Epub 2015 Apr 30. PMID 25930082